CLINICAL TRIAL: NCT00004195
Title: Evaluation of Dihydropyrimidine Dehydrogenase (DPD) Activity in Surgically Resected Primary and Metastatic Colorectal Cancer After 48 hr Pretreatment With Eniluracil
Brief Title: Eniluracil and Surgery in Treating Patients With Primary or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Glaxo Wellcome (Industry)
Responsible Party: Principal Investigator, Marty Heslin, Chief of Surgical Oncology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000067438; F980826006 (Other: University of Alabama at Birmingham IRB)
Record Dates: First submitted 2000-01-21; First posted 2004-09-16 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — eniluracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral eniluracil 20 mg twice daily (Active Comparator): 20 mg of eniluracil given twice daily for duration of the study. This subject may have surgery IF tumor is amenable to resection
  Interventions: Drug: eniluracil; Procedure: conventional colon surgery
- Placebo (Placebo Comparator): 20 mg placebo that will be given for the duration of the study. This subject may have surgery IF tumor is amenable to resection
  Interventions: Drug: eniluracil; Procedure: conventional colon surgery

INTERVENTIONS:
Drug: eniluracil — Will be given to either subject pre-operative and metastatic disease
  Other Names: 5 Fu/eniluracil (eli Lilly); 5-fu/eniluracil; 5fu/eniluraci
Procedure: conventional colon surgery — Only if the subject is amenable to surgical resections

SUMMARY:
RATIONALE: Eniluracil may increase the effectiveness of chemotherapy by blocking tumor enzymes that break down chemotherapy drugs.

PURPOSE: Randomized phase II trial to determine the effectiveness of eniluracil followed by surgery in treating patients who have primary or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the enzymatic activity of dihydropyrimidine dehydrogenase (DPD) in peripheral blood mononuclear cells (PBMC), normal mucosa, or normal liver in patients with primary or metastatic colorectal cancer. II. Evaluate the ability of eniluracil to inactivate DPD in the tumor, PBMCs, and normal tissue in this patient population. III. Assess DPD recovery and uracil levels in PBMCs following surgical resection in these patients.

OUTLINE: This is a randomized, placebo controlled study. Patients are stratified according to colorectal tumor (primary vs metastatic). Patients are randomized into one of two treatment arms. Arm I: Patients receive oral eniluracil twice daily on days -2 and -1 followed by surgical resection and tissue harvest on day 0. Arm II: Patients receive an oral placebo as in arm I followed by surgical resection and tissue harvest on day 0. Patients are followed weekly for 1 month.

PROJECTED ACCRUAL: A total of 20 patients (10 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion:

1. DISEASE CHARACTERISTICS: Histologically proven or suspicious primary or metastatic colorectal carcinoma undergoing disease resection
2. PATIENT CHARACTERISTICS:A. Age: 19 and over
3. Performance status: Karnofsky 60-100%
4. Not pregnant or nursing Fertile patients must use effective contraception during and for at least 1 month after study
5. PRIOR CONCURRENT THERAPY:
6. Subject has had at least 8 weeks since prior fluorouracil, capecitabine, fluorouracil-uracil, floxuridine, or S-1 Endocrine therapy:
7. No prior or concurrent steroids Radiotherapy:
8. Surgery: No prior emergent surgery (e.g., perforation or obstruction) No prior transplantation
9. At least 8 weeks since any prior drug metabolized by dihydropyrimidine dehydrogenase enzyme At least 8 weeks since prior flucytosine

Exclusion:

1. Severe infection(White Blood Cell Count)WBC>2 times normal
2. Fever
3. Sepsis
4. Subject on immunosuppressives therapy
5. Subjects will serum Bilirubin/Creatinine>2 times normal levels
6. Pregnant /Lactating women
7. Subjects that have received eniluracil or 5-FU(Fluorouracil) within 28 days prior to randomization
8. Subject that have comorbidity illnesses that will increase the likelihood of there death in <5 years

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1998-09; Primary Completion 1999-10 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Primary Goal to demonstrate that eniluracil at current clinical doses | Pre-operative and up to 30 days after first dose
  To see if at standard clinical doses are capable of inhibiting DPD in Primary and metastatic colorectal cancer in vivo. Since one of the mechanisms of 5-FU(Fluorouracil) tumor resistance is overexpression of DPD,effective inactivation DPD in tumors by eniluracil in this study will be supportive of the use of eniluracil to overcome this type of 5-FU(Fluorouracil) resistance

SECONDARY OUTCOMES:
Evaluate DPD recovery and uracil levels | pre-operative and up to 30 post first dose
  To evaluate the recovery of DPD and uracil levels at 4 more times in the range of postoperative days 5-7,12-16,20-24,and 26-30.

OTHER OUTCOMES:
Specific Aims | Duriation of trial up to 30 days after first dose
  1. Determine the enzymatic activity of DPD in PBMC's normal mucosa or normal liver and in primary and secondary colorectal cancers
  2. Confirm the ability of eniluracil to inactivate DPD in tumors as well as PBMC's and normal tissue
  3. Assess DPD recovery and uracil levels in PBMC's at 5-7,12-16,20-24,and 26-30 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. Heslin, MD, Study Chair — University of Alabama at Birmingham